CLINICAL TRIAL: NCT03230097
Title: A Phase II Randomised, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Orally Administered BI 409306 During a 52-week Treatment Period as an Early Intervention in Patients With Attenuated Psychosis Syndrome.
Brief Title: This Study Tests Whether BI 409306 Prevents Patients With a Specific Type of Mental Illness (Attenuated Psychosis Syndrome) From Becoming Worse. This Study Looks at How Well Patients Tolerate the Medicine and How Effective it is Over 1 Year
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: disruption due to COVID-19
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1289.32; 2016-004973-42 (EudraCT Number)
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Results first posted 2022-06-29 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders | interventions — BI 409306

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 409306 (Experimental): Patients meeting Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) diagnostic criteria for attenuated psychosis syndrome (APS) per the Structured Interview for Psychosis-Risk Syndromes (SIPS) took 50 milligrams BI 409306, as a film-coated tablet, orally twice a day at approximately the same time every day in the morning and in the evening (approximately 12 hours apart) with or without food for 52 weeks.
  Interventions: Drug: BI 409306
- Placebo (Placebo Comparator): Patients meeting Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) diagnostic criteria for attenuated psychosis syndrome (APS) per the Structured Interview for Psychosis-Risk Syndromes (SIPS) took placebo matching 50 milligrams BI 409306, as a film-coated tablet, orally twice a day at approximately the same time every day in the morning and in the evening (approximately 12 hours apart) with or without food for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 409306 — 50 milligrams BI 409306, as a film-coated tablet, orally twice a day at approximately the same time every day in the morning and in the evening (approximately 12 hours apart) with or without food for 52 weeks.
  Arms: BI 409306
Drug: Placebo — placebo matching 50 milligrams BI 409306, as a film-coated tablet, orally twice a day at approximately the same time every day in the morning and in the evening (approximately 12 hours apart) with or without food for 52 weeks.
  Arms: Placebo

SUMMARY:
This is a study in people between 16 and 30 years of age who have a specific type of mental illness called attenuated psychosis syndrome (APS). The purpose of this study is to find out whether BI 409306 helps reduce the symptoms of APS.

Participants are in the study for 1 year and 2 months. During this time, they visit the study site about 15 times and get about 10 phone calls. Participants are put into 2 groups by chance. They get either BI 409306 or placebo. Placebo tablets look like BI 409306 tablets but do not contain any medicine. Participants take a BI 409306 or placebo tablet two times a day.

During the study, participants answer questions in interviews and complete questionnaires so the doctors can check whether the APS symptoms change. The doctors also check the general health of the participants.

ELIGIBILITY:
Inclusion criteria

* Meet diagnostic criteria for attenuated psychosis syndrome as defined in DSM-5 and determined by SIPS administered at screening and diagnosis confirmed by NeuroCog Trials after review of video-taped SIPS interview.
* Age ≥16 and ≤ 30 years at the time of consent/assent.
* Male or female patients willing to use highly effective methods of contraception.

  * Female patients of childbearing potential must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. Patients must agree to use birth control throughout the trial and for at least 28 days after treatment has ended. Acceptable methods of birth control include combined estrogen-progestin oral, intravaginal or transdermal contraceptives, progestogen-only oral, injectable or implantable contraceptives, intrauterine devices (IUDs), intrauterine hormone releasing systems (IUSs), bilateral tubal occlusion, vasectomized sexual partner, and complete sexual abstinence (if acceptable by local health authorities) is allowed when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptom-thermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * Male patients who are able to father a child must be ready and able to be abstinent or use adequate contraception for the duration of study participation and for at least 28 days after treatment has ended.
* Signed and dated written informed consent in accordance with Good Clinical Practice (GCP) and local legislation prior to any study-related procedures OR signed and dated informed consent provided by the patient's parent(s) (or legal guardian) and assent by the patient prior to any study-related procedures in accordance with GCP and local legislation. If the patient has a legal representative, then this legal representative must give written informed consent as well.

Exclusion criteria

* Present or past diagnosis of schizophrenia, schizophreniform, schizoaffective disorder, bipolar disorder I, major depressive disorder with psychotic features, delusional disorder, brief psychotic disorder, other specified schizophrenia spectrum and other psychotic disorder (except attenuated psychosis syndrome), and unspecified schizophrenia spectrum and other psychotic disorder, according to DSM-5.
* Patients taking antipsychotic medication for less than 8 weeks, or patients taking antipsychotic medication for a longer duration but who have not been on a stable dose for 8 weeks prior to informed consent.
* Patients who begin taking an antipsychotic between Visit 1 and Visit 2.
* Patients who have discontinued an antipsychotic medication less than two weeks prior to randomization.
* Patients taking Clozapine.
* Suicidal behavior in the past 2 years reported in the Columbia Suicide Severity Rating Scale (C-SSRS) with a lethality of attempt ≥1, or with a lethality of 0 but a potential lethality of 2, or that in the judgement of the investigator would jeopardize the patient's safety while participating in the trial. The investigator/qualified rater must review all screening C-SSRS reports prior to randomization, documenting an additional interview assessing lethality of the behavior history when appropriate.
* Any suicidal ideation of type 4 or 5 in the Columbia Suicide Severity Rating Scale (CSSRS) in the past 3 months (i.e. active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent).
* In the judgment of the investigator, any clinically significant finding from the physical examination or laboratory value deviating from normal or any evidence of a clinically significant concomitant disease or any other clinical condition that would jeopardize a patient's safety while participating in the clinical trial.
* Known diseases of the central nervous system (including but not limited to any kind of seizures or stroke).
* History of significant head injury (>5 minutes without consciousness).
* A serious developmental disorder that in the judgement of the investigator would inhibit the patient's ability to comply with all study procedures, or mental retardation (documented IQ <70), or acute attenuated symptoms exclusively related to intoxication from a psychotropic substance.
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Planned elective surgery requiring general anesthesia, or hospitalization for more than 1 day during the study period.
* Meets criteria for Substance Use Disorder (DSM-5) within the six months prior to informed consent/assent.
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Patients taking strong or moderate CYP1A2 inhibitors who are also a CYP2C19 Poor Metabolizer (PM). Patients taking medication known to be a strong or moderate inhibitor of CYP1A2 must be prospectively genotyped to ensure they are not poor metabolizers of CYP2C19. (A list of CYP1A2 and CYP2C19 inhibitors can be found in the ISF.).
* Patients taking strong or moderate CYP1A2 inhibitors who are also taking concomitant strong or moderate CYP2C19 inhibitors. (A list of CYP1A2 and CYP2C19 inhibitors can be found in the ISF.)
* Patients with a history of moderate to severe hepatic impairment (Child-Pugh B / C).
* Patients with a history of moderate to severe renal impairment (Stage 3 - 5).
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* In the judgment of the investigator, inability of the patient to comply with the clinical trial procedures.
* Currently enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or receiving other investigational treatment(s).
* Previous participation in any BI 409306 study.
* Further exclusion criteria apply

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (33):
- United States (23):
  - ProScience Research Group, Culver City, California
  - University of California San Diego, San Diego, California
  - PRIME Clinic, New Haven, Connecticut
  - University of Florida College of Medicine, Jacksonville, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Augusta University, Augusta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - Cherry Health, Grand Rapids, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - Altea Research Institute, Las Vegas, Nevada
  - Center For Emotional Fitness, Cherry Hill, New Jersey
  - New York State Psychiatric Institute, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - PeaceHealth Medical Group, Eugene, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Community Clinical Research, Inc., Austin, Texas
  - University Hills Clinical Research, Irving, Texas
  - Psychiatric and Behavioral Solutions, LLC, Salt Lake City, Utah
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital (University of Alberta), Edmonton, Alberta
  - Chatham-Kent Clinical Trials Research Centre, Chatham, Ontario
  - Alan D. Lowe Medicine Professional Corporation, Toronto, Ontario
- China (2):
  - Peking University Sixth Hospital, Beijing
  - Shanghai Mental Health Center, Shanghai
- United Kingdom (4):
  - Holywell Hospital, Antrim
  - The Barberry National Centre for Mental Health, Birmingham
  - King's College Hospital, London
  - University of Manchester, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a "Document Sharing Agreement". For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Zhu Z, Roy D, Feng S, Vogler B. AI-based medication adherence prediction in patients with schizophrenia and attenuated psychotic disorders. Schizophr Res. 2025 Jan;275:42-51. doi: 10.1016/j.schres.2024.11.006. Epub 2024 Dec 4. PMID 39637767
- [Derived] Keefe RSE, Woods SW, Cannon TD, Ruhrmann S, Mathalon DH, McGuire P, Rosenbrock H, Daniels K, Cotton D, Roy D, Pollentier S, Sand M. A randomized Phase II trial evaluating efficacy, safety, and tolerability of oral BI 409306 in attenuated psychosis syndrome: Design and rationale. Early Interv Psychiatry. 2021 Oct;15(5):1315-1325. doi: 10.1111/eip.13083. Epub 2020 Dec 22. PMID 33354862
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, placebo-controlled, double-blind, parallel group trial over 52 weeks. The patients were randomised to 1 of the 2 treatment groups at a ratio of 1:1. After completion of the treatment period, or following early discontinuation, patients were to complete a 4-weeks follow-up period.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | BI 409306 | Placebo
Started | 24 | 26
Completed | 9 | 10
Not Completed | 15 | 16
Not completed — Adverse Event | 2 | 1
Not completed — non-compliance | 0 | 1
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Trial termination | 4 | 5
Not completed — Covid-19 pandemic outbreak | 0 | 1
Not completed — outcome event | 0 | 1

BASELINE CHARACTERISTICS:
Population: The treated set (TS) includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 409306 | Placebo | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.4 (4) | 20.9 (3.8) | 22.1 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 19 | 24 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 16 | 21 | 37
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Schizophrenia Cognition Rating Scale (SCoRS) total score [Mean (Standard Deviation); unit: Score on a scale] — Schizophrenia Cognition Rating Scale (SCoRS) total score. The SCoRS is a 20-item interview-based assessment of cognitive deficits and the degree to which they affect day-to-day functions. It collects information from a patient interview, interview with an informant (if available), and the administering clinician. Each of the 20 items of the SCoRS is rated on a 4-point scale (minimum of 1 and maximum of 4). Higher ratings reflect a greater degree of impairment. The composite score will be the sum of the 20 items (minimum of 20 and maximum of 80).
  Score on a scale | 36.333 (7.405) | 36.462 (7.814) | 36.400 (7.543)
Brief Assessment of Cognition (BAC App) composite T score [Mean (Standard Deviation); unit: T-score] — Brief Assessment of Cognition (BAC App) composite T score (averages five of the standardized scaled sub-test scores, token motor test score not included). The BACS consists of five tests assessing multiple domains of cognitive function: Verbal Memory, Digit Sequencing, Semantic and Letter Fluency, Symbol Coding, and Tower of London. A composite T score that is calculated using the five standardized scaled sub-test scores will be generated, larger T-score indicates better cognition. T-scores in the general population have a mean of 50 and standard deviation of 10.
  T-score | 52.417 (7.945) | 49.308 (13.451) | 50.800 (11.154)
Positive and Negative Syndrome Scale (PANSS) [Mean (Standard Deviation); unit: Score on a scale] — The PANSS positive and negative symptom scales each have 7 items, and the General Psychopathology Scale (not reported) has 16 items. The patient is rated from 1 to 7 on the 30 different items based on the interview, as well as reports from an informant when possible. Total score is the sum of the score of the 30 items (minimum 30, maximum 210), subtotal are the sum of either the positive or negative scales (minimum 7, maximum 49), lower scores represent an improvement in schizophrenia symptoms.
  Score on a scale
    Positive scale subtotal | 16.0 (3.9) | 14.5 (3.4) | 15.2 (3.7)
    Negative scale subtotal | 14.4 (5.1) | 13.4 (3.3) | 13.9 (4.2)
    total | 62.8 (12.5) | 58.2 (11.0) | 60.4 (11.8)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Remission From Attenuated Psychosis Syndrome (APS) Within a 52-week Timeframe
Description: Incidence of remission from attenuated psychosis syndrome (APS) within a 52-week timeframe. The incidence rate per patient-years of remission from attenuated psychosis syndrome (APS) is reported. Remission from APS is defined as a score of <3 on all of the five Positive Symptom items of the Scale of Prodromal Symptoms (SOPS) and maintained until the end of treatment. The SOPS provides a 6-point scale (minimum of 0 and maximum of 6, higher score indicating worse symptoms) to quantitatively rate the severity of five attenuated positive symptoms. incidence rate = number of events/total time at risk [patient-years].
Time Frame: Up to 52 weeks.
Population: Full Analysis Set (FAS): All patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment and who have analysable data (observed or imputed) in at least one efficacy endpoint.
Measure: Number; unit: remissions per patient-years
Arm/Group | BI 409306 | Placebo
Number analyzed (Participants) | 24 | 26
remissions per patient-years | 0.433 | 0.446
Statistical Analysis 1: Comparison: BI 409306 vs Placebo; Test type: Other; p = 0.7873, Regression, Cox; Stratified (by baseline use of antipsychotic medication) Cox proportional hazards model was used. Treatment effect and NAPLS risk score as covariates; Hazard Ratio (HR) = 0.849, 95% CI 2-sided [0.258 to 2.795] — Ratio = BI 409306/placebo

2. Secondary Outcome: Incidence of First Episode of Psychosis
Description: Incidence of first episode of psychosis. The incidence rate per patient-years of psychosis is reported, psychosis is defined as one or more positive Scale of Prodromal Symptoms (SOPS) symptoms rated a 6 AND either a symptom is seriously disorganizing or dangerous OR one of the symptoms above occurred at least one hour per day at an average frequency of four days/week over the past month. OR a new prescription or increase in dose of an ongoing antipsychotic medication. The SOPS provides a 6-point scale (minimum of 0 and maximum of 6, higher score indicating worse symptoms) to quantitatively rate the severity of five attenuated positive symptoms.
Time Frame: Up to 52 weeks.
Population: as for outcome 1
Measure: Number; unit: first episodes per patient-years
Arm/Group | BI 409306 | Placebo
Number analyzed (Participants) | 24 | 26
first episodes per patient-years | 0 | 0.125

3. Secondary Outcome: Change From Baseline in Everyday Functional Capacity as Measured by Schizophrenia Cognition Rating Scale (SCoRS) Total Score After 24 and 52 Weeks of Treatment
Description: Change from baseline (Day -28 to -7) in everyday functional capacity as measured by Schizophrenia Cognition Rating Scale (SCoRS) total score after 24 and 52 weeks of treatment. 20-item assessment of cognitive deficits and the degree to which they affect day-to-day functions. Each of the 20 items of the SCoRS is rated on a 4-point scale (minimum of 1 and maximum of 4). Higher ratings reflect a greater degree of impairment. The composite score will be the sum of the 20 items (minimum of 20 and maximum of 80). Data analyzed using the restricted maximum likelihood (REML) mixed effects model with repeated measurements (MMRM) including fixed, categorical effects of treatment, visit, treatment by visit interaction, baseline North American Prodromal Longitudinal Study (NAPLS) risk score, baseline use of antipsychotic medication and continuous fixed covariates of baseline score and baseline-by-visit interaction.
Time Frame: Baseline, week 24 and week 52.
Population: All patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment and who have analysable data (observed or imputed) for both timepoints in this endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | BI 409306 | Placebo
Number analyzed (Participants) | 10 | 15
Score on a scale
  Adjusted mean change from baseline at week 24 | -2.12 [-7.721 to 3.484] | -3.89 [-8.925 to 1.148]
  Adjusted mean change from baseline at week 52: number analyzed (Participants) | 9 | 10
  Adjusted mean change from baseline at week 52 | -3.05 [-8.881 to 2.778] | -6.23 [-11.530 to -0.927]
Statistical Analysis 1: Comparison: BI 409306 vs Placebo; BI 409306 vs. placebo of change from baseline at week 24. Restricted maximum likelihood (REML) mixed effects model with repeated measurements (MMRM) including fixed, categorical effects of treatment, visit, treatment by visit interaction, baseline North American Prodromal Longitudinal Study (NAPLS) risk score, baseline use of antipsychotic medication and continuous fixed covariates of baseline score and baseline-by-visit interaction; Test type: Other; p = 0.5212, Mixed Models Analysis; Adjusted mean difference = 1.77, 95% CI 2-sided [-3.773 to 7.315]
Statistical Analysis 2: Comparison: BI 409306 vs Placebo; BI 409306 vs. placebo of change from baseline at week 52. Restricted maximum likelihood (REML) mixed effects model with repeated measurements (MMRM) including fixed, categorical effects of treatment, visit, treatment by visit interaction, baseline North American Prodromal Longitudinal Study (NAPLS) risk score, baseline use of antipsychotic medication and continuous fixed covariates of baseline score and baseline-by-visit interaction; Test type: Other; p = 0.3127, Mixed Models Analysis; Adjusted mean difference = 3.18, 95% CI 2-sided [-3.071 to 9.425] — Restricted maximum likelihood (REML) mixed effects model with repeated measurements (MMRM), see endpoint description for details

4. Secondary Outcome: Change From Baseline in the Tablet Based Brief Assessment of Cognition (BAC App) Composite T Score After 52 Weeks of Treatment
Description: Change from baseline (Day -28 to -7) in the tablet based Brief Assessment of Cognition (BAC App) composite T score after 52 weeks of treatment. The BAC consists of five tests assessing multiple domains of cognitive function: Verbal Memory, Digit Sequencing, Semantic and Letter Fluency, Symbol Coding, and Tower of London. A composite T score that is calculated using the five standardized scaled sub-test scores was generated (averages five of the standardized scaled sub-test scores, token motor test score not included), larger T-score indicates better cognition. Data analyzed using the REML MMRM including fixed, categorical effects of treatment, visit, treatment by visit interaction, baseline North American Prodromal Longitudinal Study (NAPLS) risk score, baseline use of antipsychotic medication and continuous fixed covariates of baseline score and baseline-by-visit interaction. T-scores in the general population have a mean of 50 and standard deviation of 10.
Time Frame: Baseline and week 52.
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | BI 409306 | Placebo
Number analyzed (Participants) | 6 | 10
T-score | -1.51 [-7.950 to 4.929] | 3.48 [-1.641 to 8.597]
Statistical Analysis 1: Comparison: BI 409306 vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Other; p = 0.1602, Mixed Models Analysis; Adjusted mean difference = -4.99, 95% CI 2-sided [-12.033 to 2.057]

5. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Positive Items Score, Negative Items Score, and Total Score After 52 Weeks of Treatment
Description: Change from baseline (Day -28 to -7) in Positive and Negative Syndrome Scale (PANSS) positive items score, negative items score, and total score after 52 weeks of treatment. The PANSS positive and negative symptom scales each have 7 items, and the General Psychopathology Scale (not reported) has 16 items. The patient is rated from 1 to 7 on the 30 different items based on the interview, as well as reports from an informant when possible. Total score is the sum of the score of the 30 items (minimum 30, maximum 210), subtotal are the sum of either the positive or negative scales (minimum 7, maximum 49), lower scores represent an improvement in schizophrenia symptoms. Data analyzed using the REML MMRM including fixed, categorical effects of treatment, visit, treatment by visit interaction, baseline NAPLS risk score, baseline use of antipsychotic medication and continuous fixed covariates of baseline score and baseline-by-visit interaction.
Time Frame: Baseline and week 52.
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | BI 409306 | Placebo
Number analyzed (Participants) | 9 | 10
Score on a scale
  Adjusted mean change from baseline at week 52, positive items score | -3.83 [-6.355 to -1.296] | -3.03 [-5.312 to -0.743]
  Adjusted mean change from baseline at week 52, negative items score | -0.98 [-3.571 to 1.609] | -2.41 [-4.788 to -0.032]
  Adjusted mean change from baseline at week 52, total score | -6.02 [-14.396 to 2.360] | -7.73 [-15.216 to -0.245]
Statistical Analysis 1: Comparison: BI 409306 vs Placebo; BI 409306 vs. placebo of change from baseline at week 52, positive items score. Restricted maximum likelihood (REML) mixed effects model with repeated measurements (MMRM) including fixed, categorical effects of treatment, visit, treatment by visit interaction, baseline North American Prodromal Longitudinal Study (NAPLS) risk score, baseline use of antipsychotic medication and continuous fixed covariates of baseline score and baseline-by-visit interaction; Test type: Other; p = 0.5858, Mixed Models Analysis; Adjusted mean difference = -0.80, 95% CI 2-sided [-3.749 to 2.153]
Statistical Analysis 2: Comparison: BI 409306 vs Placebo; BI 409306 vs. placebo of change from baseline at week 52, negative items score. Restricted maximum likelihood (REML) mixed effects model with repeated measurements (MMRM) including fixed, categorical effects of treatment, visit, treatment by visit interaction, baseline North American Prodromal Longitudinal Study (NAPLS) risk score, baseline use of antipsychotic medication and continuous fixed covariates of baseline score and baseline-by-visit interaction; Test type: Other; p = 0.3445, Mixed Models Analysis; Adjusted mean difference = 1.43, 95% CI 2-sided [-1.604 to 4.462]
Statistical Analysis 3: Comparison: BI 409306 vs Placebo; BI 409306 vs. placebo of change from baseline at week 52, total score. Restricted maximum likelihood (REML) mixed effects model with repeated measurements (MMRM) including fixed, categorical effects of treatment, visit, treatment by visit interaction, baseline North American Prodromal Longitudinal Study (NAPLS) risk score, baseline use of antipsychotic medication and continuous fixed covariates of baseline score and baseline-by-visit interaction; Test type: Other; p = 0.7154, Mixed Models Analysis; Adjusted mean difference = 1.71, 95% CI 2-sided [-7.772 to 11.196]

ADVERSE EVENTS:
Time Frame: From treatment start date until the date of discontinuation of trial medication + 7 days, up to 381 days.
Description: The treated set (TS) includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Arm/Group | Placebo | BI 409306
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/26 | 1/24
Other Adverse Events (participants affected / at risk) | 16/26 | 21/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | BI 409306 (N=24)
Seizure (Nervous system disorders) | 1 | 0
Suicidal behaviour (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | BI 409306 (N=24)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Chromatopsia (Eye disorders) | 0 | 3
Dyschromatopsia (Eye disorders) | 0 | 3
Photophobia (Eye disorders) | 2 | 8
Visual impairment (Eye disorders) | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 5 | 0
Fatigue (General disorders) | 2 | 3
Pyrexia (General disorders) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 4 | 0
Weight increased (Investigations) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Dizziness (Nervous system disorders) | 1 | 8
Headache (Nervous system disorders) | 8 | 5
Anxiety (Psychiatric disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 1 | 5
Nightmare (Psychiatric disorders) | 2 | 0
Sleep disorder (Psychiatric disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
The sponsor decided to prematurely stop enrollment. This decision was based on the unfortunate inability to meet expected enrolment goals, a situation made far worse by the impact of the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT03230097/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT03230097/SAP_001.pdf